CLINICAL TRIAL: NCT01304407
Title: Evaluation of Calcium Absorption in Patients With Rothmund-Thomson Syndrome
Brief Title: Calcium Absorption in Patients With Rothmund-Thomson Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: United States Department of Agriculture (USDA) (U.S. Federal Agency); National Institutes of Health (NIH) (NIH); National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH); Gillson-Longenbaugh Foundation (Other)
Responsible Party: Principal Investigator, Steve Abrams, MD, Professor, Baylor College of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: H-27088; R01AR059063 (NIH)
Record Dates: First submitted 2011-02-23; First posted 2011-02-25 (Estimated); Results first posted 2020-07-08 (Actual); Last update posted 2020-07-23 (Actual); Status verified 2020-07

CONDITIONS: Rothmund-Thomson Syndrome
Keywords: Rothmund-Thomson Syndrome; Calcium absorption; Bone density
MeSH Terms: conditions — Rothmund-Thomson Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- RTS Subjects, Calcium Isotope (Other): Subjects consume breakfast and 180 ml of calcium-fortified orange juice to which 20 mg of 46Ca stable isotope was added. Immediately after breakfast, subjects receive 5 mg of 42Ca intravenously.
  Interventions: Other: Calcium stable isotope

INTERVENTIONS:
Other: Calcium stable isotope — Subjects consume breakfast and 180 ml of calcium-fortified orange juice to which 20 mg of 46Ca stable isotope was added. Immediately after breakfast, subjects receive 5 mg of 42Ca intravenously.

SUMMARY:
Osteosarcoma is the most common malignant bone tumor in children and adolescents. Because cure rates for osteosarcoma have remained stagnant for the past several decades despite numerous trials of chemotherapy agents, novel therapies based on the understanding of the molecular pathogenesis of osteosarcoma are needed. Rothmund-Thomson Syndrome (RTS) is a genetic disorder affecting many parts of the body and resulting in major skeletal abnormalities. This disease also has the propensity to increase the risk of developing cancer, particularly osteosarcoma. Two-thirds of RTS patients have a high risk of developing osteosarcoma. Therefore, it is important to understand the impact of RTS on the skeletal phenotype (as measured by bone density) in order to develop effective therapies to battle osteosarcoma.

DETAILED DESCRIPTION:
This is an evaluation of bone calcium deposition in patients with Rothmund-Thomson Syndrome (RTS).

This study includes one study visit during which subjects will be admitted to the inpatient unit in the Pediatric GCRC at TCH where they will undergo comprehensive clinical evaluations by a team of physicians familiar with RTS as well as bone-specific studies divided into four parts. Procedures for this study may be combined with procedures for H-9106, another protocol for patients with RTS by Dr. Wang.

Subjects will arrive at the GCRC at TCH after an overnight fast. Per TCH pain management protocols, numbing creams and sprays will be offered to the subject prior to the blood draw. Tylenol per TCH pain protocol is allowed. All food and beverages consumed at the GCRC will be pre-arranged by the study dietitian and weighed by the GCRC nutrition staff. Additional food is not allowed unless approved by the study dietitian.

Subjects will be asked to provide a 3-day written dietary history as well as food preferences for the GCRC study day. For the first meal of the study day, subjects will consume 180 mL of low-fat milk or orange juice to which 20 micrograms of 46Ca will have been added. (If milk is used as the vehicle for the isotope, the 46Ca will be added 18-24 hours in advance.)

Immediately after breakfast, subjects will receive 5 mg of 42Ca intravenously over 2-3 minutes. The beginning of this infusion will serve as Time 0. After the infusion is complete, the catheter hub will be changed in preparation for the subsequent blood draws. Samples for calcium isotope ratio measurement (0.5 ml of whole blood) will be obtained at 6, 12, 20, 40, 120, 180, 240, and 480 minutes after the infusion.

GCRC will provide weighed diets for the study day as directed by the study dietitian. Each meal should contain approximately 300 mg of calcium and each snack should provide negligible calcium. A complete 24-hour urine collection in 8 hour aliquots will be performed while at the GCRC starting with the first void after the isotopes are given.

After completion of this 24 hour period, the subjects will be discharged. They will continue to collect all of their urine in 8 hour aliquots for an additional 24 hours and then will collect three spot urine samples each day for the next 6 days. These samples will then be mailed to the CNRC research laboratory of Dr. Steven Abrams where they will be analyzed for isotope ratios by mass spectrometry analysis.

Upon discharge, subjects will receive a food scale and instruction sheets on recording their dietary intake for the next 3 days (i.e., weighed food record). While inpatient, the study dietitian will instruct the family on the guidelines for recording this intake. After the 3 days, the food scale and records will be returned to the CNRC for analysis.

ELIGIBILITY:
Inclusion Criteria:

* Patients at least four years of age who have been diagnosed clinically with RTS by a physician.

Exclusion Criteria:

* Any person who does not meet the inclusion criteria.

Min Age: 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2011-03; Primary Completion 2015-10 (Actual); Study Completion 2017-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Wang, MD, Principal Investigator — Baylor College of Medicine
Locations (1):
- Baylor College of Medicine / Texas Children's Hospital, Houston, Texas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The isotope tracer is used as a method to evaluate calcium absorption.
Groups:
- RTS Patients: Rothmond-Thompson patients receiving 5 mg 42Ca, 46Ca stable isotopes to evaluate bone calcium deposition
Period: Overall Study
Arm/Group | RTS Patients
Started | 29
Completed | 29
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | RTS Patients
Number analyzed (Participants) | 29
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 20
  Between 18 and 65 years | 9
  >=65 years | 0
Age, Continuous [Median (Full Range); unit: years] | 5 [1 to 49]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 13
Region of Enrollment [Number; unit: count of participants]
  United States | 29

OUTCOME MEASURES:

1. Primary Outcome: Bone Density (Low Areal Bone Mineral Density (aBMD))
Description: Individuals had low areal bone mineral density (aBMD) assessed by DXA using a Hologic Delphi-A instrument (Bedford, MA) at the Body Composition Laboratory of the Children's Nutrition Research Center, Houston, TX. Scans were performed of the whole body, lumbar spine, and proximal femur. Bone mineral content (BMC), bone area, and BMD were measured using Hologic Discovery V12.1 analysis software. For adult subjects, BMD Z-scores of the whole body, lumbar spine, left total hip, and left femoral neck were calculated using the Hologic Reference Database. Validated age- and sex-matched control data from the pediatric population generated by the Body Composition Laboratory of the Children's Nutrition Research Center, Houston, TX were used to calculate the Z-scores for pediatric subjects as previously published.
Time Frame: 8 days
Population: Areal bone mineral density (aBMD) z-scores of 13 pediatric patients, 9 adult patients. 7 of the patients did not have successful bone density scans to be included in the analysis.
Measure: Median (Inter-Quartile Range); unit: z-score
Arm/Group | RTS Patients
Number analyzed (Participants) | 22
z-score
  13 pediatric patients, whole body aBMD: number analyzed (Participants) | 13
  13 pediatric patients, whole body aBMD | -1.3 [-1.6 to -0.4]
  9 adult patients, whole body aBMD: number analyzed (Participants) | 9
  9 adult patients, whole body aBMD | -0.9 [-1.2 to 0.94]
  13 pediatric patients, lumbar spine aBMD: number analyzed (Participants) | 13
  13 pediatric patients, lumbar spine aBMD | -2.4 [-2.9 to -1.7]
  9 adult patients, lumbar spine aBMD: number analyzed (Participants) | 9
  9 adult patients, lumbar spine aBMD | -1.2 [-1.8 to 0.1]
  13 pediatric patients, femoral neck aBMD: number analyzed (Participants) | 13
  13 pediatric patients, femoral neck aBMD | -2.4 [-3.3 to -1.1]
  9 adult patients, femoral neck aBMD: number analyzed (Participants) | 9
  9 adult patients, femoral neck aBMD | -0.8 [-1.5 to 0.3]
  13 pediatric patients, total hip aBMD: number analyzed (Participants) | 13
  13 pediatric patients, total hip aBMD | -1.5 [-2.4 to -0.2]
  9 adult patients, total hip aBMD: number analyzed (Participants) | 9
  9 adult patients, total hip aBMD | -0.7 [-1.5 to 0.1]

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | RTS Patients
All-Cause Mortality (participants affected / at risk) | 0/29
Serious Adverse Events (participants affected / at risk) | 0/29
Other Adverse Events (participants affected / at risk) | 0/29

LIMITATIONS AND CAVEATS:
Single measurement of bone density is less informative than serial measurements. Individuals with RTS are typically below the 5th percentile for height, and thus age adjusted Z-scores may overestimate the magnitude of low bone mass.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No